CLINICAL TRIAL: NCT01209351
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dosing, Parallel Group Study to Assess the Effects of Teduglutide (ALX-0600) on Gastric Emptying in Healthy Subjects
Brief Title: Effect of Teduglutide on Gastric Emptying in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: C10-003
Record Dates: First submitted 2010-09-20; First posted 2010-09-27 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Pharmacodynamics; teduglutide
MeSH Terms: interventions — teduglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- teduglutide (Experimental)
  Interventions: Drug: teduglutide

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: Placebo
Drug: teduglutide — teduglutide 4 mg
  Arms: teduglutide

SUMMARY:
The primary objective of this study is to assess the effects of 10 consecutive, daily, subcutaneous doses of 4 mg of teduglutide as compared with placebo on gastric emptying as assessed by acetaminophen absorption kinetics in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the nature of the study and have agreed to and are able to read, review, understand, and sign the informed consent document prior to any screening assessments being completed.
2. Completed the screening process within 30 days prior to check in
3. Adult males or females age 18 to 45 years in good health as determined by medical history, physical examination, ECG, and laboratory tests
4. Women who are: (1) post-menopausal; (2) surgically sterilized, OR (3) of childbearing potential with a negative pregnancy test at screening and check-in and who consent to use an acceptable method of contraception for the duration of the study and for four weeks following last dose of study drug.

Exclusion Criteria:

1. Allergy or sensitivity to acetaminophen
2. History of structural abnormality or pathology of the GI tract or diseases/conditions which affect GI motility including the following:

Gastric, small bowel or colonic resection, Colon cancer or any GI Tract cancer Inflammatory bowel disease, Irritable bowel disease, Diabetes Mellitus, Gallstones or cholecystectomy, Appendectomy, hernia repair, benign polypectomy are not excluded, History of Gilbert's Syndrome 3 History of hepatitis or pancreatitis 4 Evidence of any abnormal hepatobiliary laboratory parameters (> ULN for serum ALT; AST; ALP; GGT; and/or total, direct or indirect bilirubin) 5 Serum amylase or lipase above the upper limit of normal 6 Body mass index (BMI) > 30 kg/m2 7 Intention to use medication that potentially affects GI tract motility 8 History of a viral or bacterial infection, allergy, other inflammatory process or surgery within 3 weeks of the check-in day.

9 Clinical evidence or history (including that from medical and medication history, physical examination, laboratory, ECG and any other available test results such as those from medical imaging studies) of significant cardiovascular, respiratory, renal, gastrointestinal, hematologic (eg, anemia), neurologic, psychiatric conditions or of any disease that may interfere with the objectives of the study or with the subject successfully completing the study 10 Presently taking prescription or over the counter medication including products containing acetaminophen, vitamins, herbs or dietary supplements, which cannot be discontinued. Prohibited medications must be discontinued at least 7 days prior to check-in and all other medications and supplements must be stopped at least 72 hours prior to check-in.

11 Current or recent history (within 12 months) of drug or alcohol abuse 12 Positive drug or alcohol screen 13 Current or recent history (within 3 months) of use of tobacco products 14 Positive urine cotinine screen 15 Abnormalities in clinical chemistry, hematology, urinalysis or in any other laboratory variables 16 Positive results in any of the virology tests of acute or chronic infectious human immunodeficiency virus (HIV) and hepatitis virus infections 17 Pregnant or lactating females; positive beta human chorionic gonadotropin (b-hCG) pregnancy test in females only 18 Special dietary requirements which would preclude a subject's acceptance of a high fat or high caloric, standardized meal 19 Blood donation within 4 weeks of the check-in day 20 Participation in another clinical trial with an investigational drug or device within the last month (if single dose) and at least 3 months (if multiple dose) or within 10 times the half-life of the respective investigational drug, whatever is longer, before the screening evaluation. For biologics the minimum period is at least 6 months or the time of duration of the pharmacodynamic effect or 10 times the half-life of the respective drug, whatever is longer, before the screening evaluation.

21 Lack of ability or willingness to give informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09-28 (Actual); Primary Completion 2010-11-08 (Actual); Study Completion 2010-11-08 (Actual)

PRIMARY OUTCOMES:
PK log-transformed parameters AUC and CMax | Day 10
  The primary objective of this study is to assess the effects of 10 consecutive, daily, subcutaneous doses of 4 mg of teduglutide as compared with placebo on gastric emptying as assessed by acetaminophen absorption kinetics in healthy subjects.

SECONDARY OUTCOMES:
AUC for each GI blood markers | day 10
  The secondary objectives of this study are to assess the effects of subcutaneous dosing of 4 mg of teduglutide administered in single daily doses on the pharmacokinetics of teduglutide on the AUC 3 hours post dose on insulin, glucose, and glucagon.
CMax | Day 10
  The secondary objectives of this study are to assess the effects of subcutaneous dosing of 4 mg of teduglutide administered in single daily doses on the pharmacokinetics of teduglutide on the cMax 3 hours post dose on insulin, glucose, and glucagon.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Cetero Clinical Research, San Antonio, Texas, United States

REFERENCES:
- [Derived] Berg JK, Kim EH, Li B, Joelsson B, Youssef NN. A randomized, double-blind, placebo-controlled, multiple-dose, parallel-group clinical trial to assess the effects of teduglutide on gastric emptying of liquids in healthy subjects. BMC Gastroenterol. 2014 Feb 12;14:25. doi: 10.1186/1471-230X-14-25. PMID 24517114